CLINICAL TRIAL: NCT01170091
Title: Safety and Effect of Mirapex(Pramipexole) Tablet Among Korean RLS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.653
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pramipexole

SUMMARY:
Safety and Effect of Mirapex(Pramipexole) tablet among Korean Restless Legs Syndrome Patients: An Open-Label, Postmarketing Surveillance Study

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Moderate to severe Primary Restless Legs Syndrome
2. Male or female patients aged at least 18 years

Exclusion criteria:

1. Any contraindications according to Basic Product Information (Company Core Data Sheet) or local Labelling; hypersensitivity to pramipexole or to any of the excipients.
2. Ongoing treatment with Mirapex
3. Pregnant and breastfeeding women
4. Concomitant pharmacologic treatment with other dopaminergic drugs(including L-dopa)
5. Secondary RLS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General hospitals, primary care clinics
Sampling Method: Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2007-12; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- South Korea (36):
  - Boehringer Ingelheim Investigational Site 1, Busan
  - Boehringer Ingelheim Investigational Site 2, Busan
  - Boehringer Ingelheim Investigational Site 3, Busan
  - Boehringer Ingelheim Investigational Site 32, Daegu
  - Boehringer Ingelheim Investigational Site 33, Daegu
  - Boehringer Ingelheim Investigational Site 34, Daejeon
  - Boehringer Ingelheim Investigational Site 35, Daejeon
  - Boehringer Ingelheim Investigational Site 36, Deajeon
  - Boehringer Ingelheim Investigational Site 25, Gwangju
  - Boehringer Ingelheim Investigational Site 26, Gwangju
  - Boehringer Ingelheim Investigational Site 27, Gwangju
  - Boehringer Ingelheim Investigational Site 28, Gwangju
  - Boehringer Ingelheim Investigational Site 29, Gwangju
  - Boehringer Ingelheim Investigational Site 30, Gwangju
  - Boehringer Ingelheim Investigational Site 31, Gwangju
  - Boehringer Ingelheim Investigational Site 10, Seoul
  - Boehringer Ingelheim Investigational Site 11, Seoul
  - Boehringer Ingelheim Investigational Site 12, Seoul
  - Boehringer Ingelheim Investigational Site 13, Seoul
  - Boehringer Ingelheim Investigational Site 14, Seoul
  - Boehringer Ingelheim Investigational Site 15, Seoul
  - Boehringer Ingelheim Investigational Site 16, Seoul
  - Boehringer Ingelheim Investigational Site 17, Seoul
  - Boehringer Ingelheim Investigational Site 18, Seoul
  - Boehringer Ingelheim Investigational Site 19, Seoul
  - Boehringer Ingelheim Investigational Site 20, Seoul
  - Boehringer Ingelheim Investigational Site 21, Seoul
  - Boehringer Ingelheim Investigational Site 22, Seoul
  - Boehringer Ingelheim Investigational Site 23, Seoul
  - Boehringer Ingelheim Investigational Site 24, Seoul
  - Boehringer Ingelheim Investigational Site 4, Seoul
  - Boehringer Ingelheim Investigational Site 5, Seoul
  - Boehringer Ingelheim Investigational Site 6, Seoul
  - Boehringer Ingelheim Investigational Site 7, Seoul
  - Boehringer Ingelheim Investigational Site 8, Seoul
  - Boehringer Ingelheim Investigational Site 9, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirapex: Patients with RLS who had initiated with Mirapex
Period: Overall Study
Arm/Group | Mirapex
Started | 651
Completed | 627
Not Completed | 24
Not completed — Missing efficacy evaluation | 3
Not completed — Treatment duration is less than 4 weeks | 21

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Patients With Restless Legs Syndrome (RLS): Patients with RLS who had initiated with Mirapex
Arm/Group | Patients With Restless Legs Syndrome (RLS)
Number analyzed (Participants) | 651
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (13.2)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 369
  Male | 276
  Not reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Adverse Events
Description: If there is a dose titration, another 4 weeks should be followed up
Time Frame: Up to 4 weeks
Population: Patients with RLS who took at least one dose of Mirapex - Safety Analysis Set
Measure: Number; unit: cases
Arm/Group | Mirapex
Number analyzed (Participants) | 651
cases
  Gastrointestinal disorders | 8
  Nervous system disorders | 1
  General disorders and admin site conditions | 2
  Psychiatric disorders | 1

2. Secondary Outcome: International Restless Legs Syndrome Rating Scale (IRLS) Change After 4 Weeks of Mirapex Treatment
Description: a change in 10-item scale rated by the patient on 5 levels with a minimum ("none") sum score of 0 to maximum ("very severe") sum score of 40
Time Frame: before and after the treatment with Mirapex (at least 4 weeks after the end of titration)
Population: Patients whose IRLS scores were assessed at the baseline and at 4 weeks after the end of titration. Efficacy data set (Intent to Treat)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Mirapex
Number analyzed (Participants) | 627
Units on a scale | -14.7 (7.6)

3. Secondary Outcome: Patient-Global Impressions (PGI-I)
Description: PGI comprises of 7 categories including "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse" and "very much worse."
Time Frame: before and after the treatment with Mirapex (at least 4 weeks after the end of titration)
Population: Patients whose PGI were assessed at the baseline and at 4 weeks after the end of titration. Efficacy Data Set (Intent to Treat)
Measure: Number; unit: patients
Arm/Group | Mirapex
Number analyzed (Participants) | 627
patients
  Very much improved | 177
  Much improved | 360
  Minimally improved | 45
  No change | 42
  Minimally worse | 2
  Much worse | 1
  Very much worse | 0

4. Secondary Outcome: Clinical Global Impressions-Global Improvement (CGI-I)
Description: CGI-I comprises of 7 categories including "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse" and "very much worse."
Time Frame: before and after the treatment with Mirapex (at least 4 weeks after the end of titration)
Population: Patients whose CGI-I were assessed at the baseline and at 4 weeks after the end of titration. Efficacy Data Set (Intent to Treat)
Measure: Number; unit: patients
Arm/Group | Mirapex
Number analyzed (Participants) | 627
patients
  Very much improved | 188
  Much improved | 351
  Minimally improved | 49
  No change | 35
  Minimally worse | 3
  Much worse | 1
  Very much worse | 0

ADVERSE EVENTS:
Time Frame: 4 weeks (28 days)
Arm/Group | Patients With Restless Legs Syndrome (RLS)
Serious Adverse Events (participants affected / at risk) | 0/651
Other Adverse Events (participants affected / at risk) | 0/651

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.